CLINICAL TRIAL: NCT04331236
Title: Yoga-Cognitive Behavioral Therapy (Y-CBT) Group Intervention for Adolescents With Chronic Pain and Their Caregivers: A Feasibility Study
Brief Title: Yoga-CBT Group Intervention for Adolescents With Chronic Pain and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-015337
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Chronic Pain
Keywords: pediatric pain; cognitive behavioral therapy; yoga
MeSH Terms: interventions — Cognitive Behavioral Therapy; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient and Caregiver Intervention (Experimental): Patient and Caregivers receive both cognitive behavioral intervention and yoga interventions each week, for 7 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Other: Yoga

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT trains individuals to identify and reframe dysfunctional thoughts to help improve mood and behavior. CBT intervention also includes teaching relaxation and mindfulness strategies, as well as ways to help improve functioning through the use of behavioral goal setting.
Other: Yoga — Yoga consists of physical exercises, breathing techniques, and meditation designed to condition the physical body, calm the mind, and stabilize emotions.

SUMMARY:
Clinical symptoms that are often found to be comorbid with pediatric chronic pain include anxiety, depression as well as increased stress, obesity, and decreased physical conditioning. Integrative therapies have been increasingly offered at children's hospitals as part of an integrated approach to treatment. Limited research exits on the efficacy of mind-body practices (e.g., yoga) utilized in conjunction with evidenced-based non-pharmacological treatments like cognitive behavioral therapy (CBT) to treat pediatric pain. Hence, this 7-week interventional pilot study was conducted to evaluate the impact of combining yoga and CBT for both pediatric patients with chronic pain and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Established Children's Hospital of Philadelphia (CHOP) patients 14-18 years old, of any gender, race, or ethnicity
* English speaking
* Has received a diagnosis related to the primary symptom of chronic pain
* For adolescents who are less than 18 y/o, parental or guardian permission (informed consent) and adolescent assent (patient)
* Parents or legal guardians of adolescents enrolled, who speak English
* Parents or legal guardians' permission (informed consent) of their own participation

Exclusion Criteria:

* Current medical status or cognitive functioning precludes completing assessment instruments (e.g., cognitive or intellectual disability such as diagnosis of autism spectrum disorder)
* Physical limitation, handicap, or injury that would prevent participation or risk further injury or harm (e.g. physical assistance required from a device)
* Non-English speaking
* For adolescents who are less than 18 years of age, parental or guardian permission (informed consent) and/or adolescent (patient) assent declined
* Patient, who in the opinion of the investigator, may be non-compliant or unable to complete the study procedures
* Parents or legal guardians of adolescents enrolled, who do not speak English
* Parents or legal guardians' permission (informed consent) for their own participation or if the adolescent is less than 18 years of age and assent has been declined
* Parents or legal guardians, who in the opinion of the investigator, may be non-compliant or unable to complete the study procedures (If the dyad or triad includes a primary caregiver who has a developmental delay, intellectual disability, or communication challenge that prohibits completion of questionnaires or participation in study sessions)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Assessment of the feasibility of conducting a 7-week group intervention combining yoga and cognitive behavioral therapy (CBT) | Feasibility Questionnaires given after the 7-week intervention
  Likert-scale used to quantify satisfaction with the intervention; content clarity; concept-applicability to current life; impression of program design; scheduling considerations and other open-ended questions about their study preferences

SECONDARY OUTCOMES:
Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Pain Interference | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  Consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
PROMIS Social Health - Peer Relationships | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  Quality of relationships with friends and other acquaintances.
PROMIS Emotional Distress - Depressive Symptoms | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  Negative mood (sadness, guilt), views of self (self- criticism,worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose).
PROMIS Pediatric Global Health 7+2 | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  Overall evaluation of one's physical and mental health.
Pain Stages of Change Questionnaire - Child Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  Validated 30-item self-report measure (ages 12-18) that will assess the readiness or receptiveness of adolescents and their parents to adopt a self-management approach to pain
Pain Catastrophizing Scale - Child Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A 13-item self-report scale (ages 8-17) with versions that will evaluate catastrophizing thinking in the adolescent subjects as well as parents (in relation to their child's pain)
Adult's Responses to Children's Symptoms - Child Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A 29-item validated measure (ages 8-18) that will assess the behavior of parents (caregivers) in response to their child's pain, as self-reported by the parent (or reported by the child)
Visual Analog Pain Score | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  An established patient-reported measure that will quantify each adolescent subject's pain severity. With anchors at 0 (No pain) and 100 (Worst pain possible), these subjects will indicate the level of pain intensity on a 100 mm line
Pain Stages of Change Questionnaire - Parent Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A validated 30-item self-report measure (ages 12-18) that will assess the readiness or receptiveness of adolescents and their parents to adopt a self-management approach to pain
Pain Catastrophizing Scale - Parent Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A 13-item self-report scale (ages 8-17) with versions that will evaluate catastrophizing thinking in the adolescent subjects as well as parents (in relation to their child's pain)
Adult's Responses to Children's Symptoms - Parent Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A 29-item validated measure (ages 8-18) that will assess the behavior of parents (caregivers) in response to their child's pain, as self-reported by the parent (or reported by the child)
Brief Symptoms Inventory - Parent Proxy | Given before the intervention (Week 1), after the intervention (Week 7) and 3 months post-intervention
  A 53-item self-report measure that will assesses psychological functioning in adults. The instrument has three global indices as well as nine symptom dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hainsworth KR, Salamon KS, Khan KA, Mascarenhas B, Davies WH, Weisman SJ. A pilot study of yoga for chronic headaches in youth: promise amidst challenges. Pain Manag Nurs. 2014 Jun;15(2):490-8. doi: 10.1016/j.pmn.2012.12.002. Epub 2013 Feb 19. PMID 23428497
- [Background] Eccleston C, Palermo TM, Williams AC, Lewandowski Holley A, Morley S, Fisher E, Law E. Psychological therapies for the management of chronic and recurrent pain in children and adolescents. Cochrane Database Syst Rev. 2014 May 5;2014(5):CD003968. doi: 10.1002/14651858.CD003968.pub4. PMID 24796681
- [Background] Khalsa MK, Greiner-Ferris JM, Hofmann SG, Khalsa SB. Yoga-enhanced cognitive behavioural therapy (Y-CBT) for anxiety management: a pilot study. Clin Psychol Psychother. 2015 Jul-Aug;22(4):364-71. doi: 10.1002/cpp.1902. Epub 2014 May 7. PMID 24804619